CLINICAL TRIAL: NCT03791138
Title: The Impact of a Web-based Decision Aid for Women Considering Breast Reconstruction: a Randomized Controlled Trial
Brief Title: The Impact of a Web-based Patient Decision Aid for Women Considering Breast Reconstruction
Acronym: TANGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NKI 2014-7031; A6C/NKI 2014-7031 (Other Grant/Funding Number: Dutch Cancer Society)
Record Dates: First submitted 2018-12-17; First posted 2019-01-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; patient decision aid; decisional conflict; randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Care as usual and an online patient decision aid
  Interventions: Other: online patient decision aid
- control group (No Intervention): Care as usual with a standard information leaflet

INTERVENTIONS:
Other: online patient decision aid — An online, interactive tool that can be used to prepare for consultation with a plastic surgeon which contains evidence-based information about breast reconstruction options, the pros and cons of the options, value clarification exercises and patient narratives. It results in a summary sheet with patients' personal values and questions that can be discussed during consultation with a plastic surgeon.
  Other Names: Breast Reconstruction Decision Aid
  Arms: intervention group

SUMMARY:
This study evaluates the impact of an online patient decision aid on the process of decision making regarding breast reconstruction and the decision quality in women with breast cancer undergoing mastectomy and considering immediate breast reconstruction. Half of participants will receive care as usual and access to the online decision aid, while the other half will receive care as usual including a standard information leaflet.

DETAILED DESCRIPTION:
Rationale: In the Netherlands, of the approximately 15,000 women who are diagnosed with breast cancer each year, about 40% undergo mastectomy. A wide variety of breast reconstructive methods are offered to these women. In most cases, there is no clear medical recommendation on which procedure is the best. Decisions for breast surgery and reconstruction are frequently made during an emotionally burdensome and restricted timeframe. Women may find it hard to make a decision for the type of surgery and reconstruction, some feel that the decision is hurried and uninformed, and many have some degree of regret about their decision at a later date. To support women in making a well-informed decision about breast reconstruction, an online patient decision aid (pDA) has been developed.

Objective: The primary objective of the study is to evaluate the impact of the use of the online pDA on the process of decision making regarding breast reconstruction and the decision quality. The secondary objective of the study is to evaluate the impact of the use of the online pDA on patient reported health outcomes, to identify possible moderators of the effect, and to investigate the cost-effectiveness.

Hypotheses: It is hypothesized that the online pDA, as compared to usual care, will improve the decision making process about breast reconstruction (i.e. leads to less decisional conflict, higher satisfaction with information, higher levels of preparedness for decision making and higher perceived levels of shared decision making) and that it will improve the decision quality (i.e. leads to higher levels of knowledge about breast reconstruction and lower levels of regret).

Study design: A multicenter randomized controlled trial (RCT) will be performed in eight hospitals. All consenting participants will be randomized into one of the two study arms (intervention group or control group). Women in both groups will be invited to complete questionnaires at baseline (i.e. before randomization), 1 week after consultation with a plastic surgeon and 3 and 12 months after breast surgery.

Study population: 250 women will participate.

ELIGIBILITY:
Inclusion Criteria:

* female (≥18 years);
* diagnosed with breast cancer or carcinoma in situ;
* will be treated with mastectomy and is eligible for immediate breast reconstruction;
* is referred to a plastic surgeon (consultation takes place ≥3 working days after study invitation);
* has internet access and sufficient computer skills;
* is able to read and speak the Dutch language.

Exclusion Criteria: None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
decisional conflict | 1 week after consultation with a plastic surgeon (T1)
  decisional conflict scale (DCS); the DCS consists of a total score and five subscales (uncertainty, feeling informed, feeling clear about values, feeling supported and effective decision-making). It consists of 16 items which are rated on a 5-point Likert-type scale (strongly agree- strongly disagree). Scores range from 0 - 100, with higher scores indicating more decisional conflict.

SECONDARY OUTCOMES:
decisional conflict | 3 months after surgery (T2); 12 months after surgery (T3)
  decisional conflict scale (DCS); the DCS consists of a total score and five subscales (uncertainty, feeling informed, feeling clear about values, feeling supported and effective decision-making). It consists of 16 items which are rated on a 5-point Likert-type scale (strongly agree- strongly disagree). Scores range from 0 - 100, with higher scores indicating more decisional conflict.
decision regret | 3 months after surgery (T2); 12 months after surgery (T3)
  decision regret scale (DRS); the DRS consists of 5 items, rated on a 5 point Likert-type scale (strongly agree - strongly disagree). Scores range from 0 - 100, with higher scores indicating higher levels of regret.
knowledge about breast reconstruction | 1 week after consultation with plastic surgeon (T1); 3 months after surgery (T2); 12 months after surgery (T3)
  study-specific questionnaire consisting of 10 items (true/false/I don't know)
preparedness for decision making | 1 week after consultation with a plastic surgeon (T1)
  preparation for decision making scale; 10 items, rated on a 5-point Likert-type scale (Not at all - a great deal). Scores range from 0 - 100, with higher scores indicating higher perceived level of preparation for decision making.
satisfaction with information | 1 week after consultation with plastic surgeon (T1); 3 months after surgery (T2); 12 months after surgery (T3)
  three study-specific questions (a. How satisfied are you with the information about breast reconstruction? (5 point Likert-scale: not at all - very satisfied), b. Did you miss information? (yes/no), and c. Would you have preferred less information? (yes/no)). The subsample of women who opted for breast reconstruction will also complete the Satisfaction with Information-subscale of the Breast-Q (14 items, 4 point Likert-type scale, very dissatisfied - very satisfied, scores range from 0 -100, with higher scores indicating higher levels of satisfaction with information).
patient's perception of shared decision making | 1 week after consultation with a plastic surgeon (T1)
  shared decision making questionnaire (SDM-Q-9); the SDM-Q-9 consists of 9 items, rated on a 6 point Likert-type scale (completely disagree - completely agree). The sum of all items (score between 0 - 45) will be multiplied by 20/9 to transform scores to range from 0 -100, where 0 indicates the lowest possible level of shared decision making and 100 indicates the highest extent of shared decision making.
satisfaction with plastic surgeon | 1 week after consultation with plastic surgeon (T1)
  The subscale Satisfaction with Surgeon of the Breast-Q consists of 12 items, rated on a 4 point Likert-type scale (completely disagree - completely agree). Scores range from 0 - 100.
actual choice | 3 months after surgery (T2); 12 months after surgery (T3)
  actual choice about breast reconstruction (self-reported and verified against patients' medical records)
satisfaction with outcome | 3 months after surgery (T2); 12 months after surgery (T3)
  The Breast-Q subscale Satisfaction with Breast measures body image in terms of a woman's satisfaction with her breasts. It consists of 4 to 16 items (depending on the type of surgery), rated on a 4 point Likert-type scale (very dissatisfied - very satisfied). The subsample of women who opted for breast reconstruction also completes the Breast-Q subscale Satisfaction with Breast Outcome (7 items, 3 point Likert-type scale (disagree - completely agree)), measuring a woman's overall appraisal of the outcome of her breast surgery. For both subscales, scores range from 0 -100, with higher scores indicating higher satisfaction.
body image | 3 months after surgery (T2); 12 months after surgery (T3)
  Subscale Body Image of the EORTC QLQ-BR23 (4 items, 4 point likert-type scale (not at all - very much), scores range from: 0-100 , a higher score is better.
sexual functioning | 3 months after surgery (T2); 12 months after surgery (T3)
  Subscales of Sexual Functioning (2 items) and Sexual Enjoyment (1 item) of the EORTC-QLQ BR23. Both subscale are rated on a 4 point Likert-type scale (not at all - very much). Scores range from 0-100, a higher score is better.
breast symptoms | 3 months after surgery (T2); 12 months after surgery (T3)
  Subscale Breast Symptoms (4 items, 4 point Likert-type scale, not at all - very much) of the EORTC QLQ-BR23. Scores range from 0-100, a higher score is worse.
anxiety | 1 week after consultation with a plastic surgeon (T1); 3 months after surgery (T2); 12 months after surgery (T3)
  The short-form of the state scale of the spielberger state-trait anxiety inventory (STAI), consisting of 6 items, rated on a 4 point Likert-type scale (not at all - very much). Scores range from 20 - 80, with higher scores indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Eveline MA Bleiker, Professor, Principal Investigator — The Netherlands Cancer Institute
Locations (8):
- Netherlands (8):
  - Meander Medical Center, Amersfoort
  - Medical Center Slotervaart, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Medical Center Leeuwarden, Leeuwarden
  - Erasmus Medical Center, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ter Stege JA, Woerdeman LAE, Kieffer JM, Sherman KA, Agelink van Rentergem JA, van Duijnhoven FH, van Huizum MA, Gerritsma MA, Kuenen M, Corten EML, Kimmings NAN, Ruhe QPQ, Krabbe-Timmerman IS, Van't Riet M, Hahn DEE, Witkamp AJ, Oldenburg HSA, Bleiker EMA. Efficacy of a Decision Aid in Breast Cancer Patients Considering Immediate Reconstruction: Results of a Randomized Controlled Trial. Plast Reconstr Surg. 2024 Oct 1;154(4):706-722. doi: 10.1097/PRS.0000000000011100. Epub 2023 Oct 9. PMID 37815283
- [Derived] Ter Stege JA, Woerdeman LAE, Hahn DEE, van Huizum MA, van Duijnhoven FH, Kieffer JM, Retel VP, Sherman KA, Witkamp AJ, Oldenburg HSA, Bleiker EMA. The impact of an online patient decision aid for women with breast cancer considering immediate breast reconstruction: study protocol of a multicenter randomized controlled trial. BMC Med Inform Decis Mak. 2019 Aug 19;19(1):165. doi: 10.1186/s12911-019-0873-1. PMID 31426772